CLINICAL TRIAL: NCT03741985
Title: Effect of Dumbbell Exercise on Arteriovenous Fistula in Patients With Hemodialysis：A Prospective Randomized,Controlled Trial
Brief Title: Effect of Dumbbell Exercise on Arteriovenous Fistula in Patients With Hemodialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GDREC2016329H
Record Dates: First submitted 2018-10-28; First posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-09

CONDITIONS: Arteriovenous Fistula
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The handgrip exercise (Placebo Comparator): Patients are asked to squeeze a rubber ring 30 times per min for altogether 20 minutes on non-dialysis days.The 20-minute exercise can be divided into 3 parts according to individual circumstances.
  Interventions: Behavioral: The handgrip exercise
- The dumbbell exercise (Experimental): Patients are asked to hold 6-pound dumbbells to exercise 30 times per min for altogether 20 minutes on non-dialysis days.The 20-minute exercise can be divided into 3 parts according to individual circumstances.
  Interventions: Behavioral: The dumbbell exercise

INTERVENTIONS:
Behavioral: The handgrip exercise — The control group was given routine dialysis treatment and daily handgrip exercise .Patients are asked to squeeze a rubber ring 30 times per min for altogether 20 minutes on non-dialysis days.The 20-minute exercise can be divided into 3 parts according to individual circumstances.
  Arms: The handgrip exercise
Behavioral: The dumbbell exercise — The experimental group was given routine dialysis treatment and daily dumbbell exercise .Patients are asked to hold 6-pound dumbbells to exercise 30 times per min for altogether 20 minutes on non-dialysis days.The 20-minute exercise can be divided into 3 parts according to individual circumstances.
  Arms: The dumbbell exercise

SUMMARY:
Isometric exercise has been shown to increase the diameter and the blood flow rate of forearm veins.At present, more studies focus on the perioperative period to promote the maturation of arteriovenous fistula(AVF), while there are few reports on functional maintenance measures for the patients with maintenance hemodialysis.This study aims to explore the effect of dumbbell exercise on AVF，and evaluate whether patients can carry a 6-pound item with the fistula limb in a reasonable way.

DETAILED DESCRIPTION:
Autologous arteriovenous fistula (AVF) is the preferred vascular access for maintenance hemodialysis patients. It is estimated that AVF accounts for 85-90% of the permanent vascular access in Chinese hemodialysis patients. With the prolongation of dialysis time, aging, and the increase of diabetes incidence, the complications of AVF are more and more common, which affect the lifetime of AVF. Therefore,self-maintenance of AVF is essential. Among them, exercise should be used throughout the entire process of AVF use for the reason that it is economical, easy to operate, and highly repeatable.The most common isometric exercise is handgrip exercise. However, there are some deficiencies in this exercise, such as lack of quantitative standards and burnout of repeated actions. As a result, this study uses quantitative dumbbells as a training tool to explore the effect of dumbbell exercise on the maintenance of AVF, and further evaluates and breaks the nursing routine of "no lifting weights" of fistula limb.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have established arteriovenous fistula
2. Patients whose muscle strength of the fistula limb is graded 4-5, which can overcome the 6-pound gravity and external resistance to complete the range of joint activity
3. Patients who provided informed consent.

Exclusion Criteria:

1. Left ventricular cardiac ejection fraction <30%;
2. Using a arteriovenous graft or a long-term catheter as a permanent access;
3. The diameter of the aneurysm is greater than 2 cm or the aneurysm has a risk of rupture;
4. Participation in other clinical trials at the same time;
5. Severe cardiovascular diseases and other organ complications,malignant tumors, mental illnesses, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-11-10 (Estimated); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Changes in blood flow of AVF draining vein | from Baseline to 3 months
  The blood flow measurement was repeated three times at a location 5 cm proximal to the anastomosis in the draining vein by Doppler ultrasound.

SECONDARY OUTCOMES:
Changes in diameter of AVF draining vein | from Baseline to 3 months
  The diameter measurement was repeated three times at a location 5 cm proximal to the anastomosis in the draining vein by Doppler ultrasound.
The ratio of pre-pump arterial pressure and blood flow | from Baseline to 3 months
  The ratio of pre-pump arterial pressure and blood flow during the hemodialysis treatment.
Adverse event | from Baseline to 3 months
  The incidence of adverse event(puncture site hematoma,hemorrhage,aneurysm,heart failure,joint sprain,falls,anastomotic rupture,etc).
Changes in blood flow of AVF proximal artery | from Baseline to 3 months
  The blood flow measurement was repeated three times at a location 5 cm proximal to the anastomosis in the proximal artery by Doppler ultrasound.
Changes in blood flow of brachial artery | from Baseline to 3 months
  The blood flow measurement was repeated three times at a location 2 cm above the elbow in the brachial artery by Doppler ultrasound.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nantakool S, Reanpang T, Prasannarong M, Pongtam S, Rerkasem K. Upper limb exercise for arteriovenous fistula maturation in people requiring permanent haemodialysis access. Cochrane Database Syst Rev. 2022 Oct 3;10(10):CD013327. doi: 10.1002/14651858.CD013327.pub2. PMID 36184076